CLINICAL TRIAL: NCT00002670
Title: Phase III Intergroup Trial of Surgery Followed by (1) Radiotherapy vs. (2) Radiochemotherapy For Resectable High Risk Squamous Cell Carcinoma of the Head and Neck
Brief Title: Radiation Therapy With or Without Chemotherapy in Treating Patients With Head and Neck Cancer That Has Been Removed During Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9501; CDR0000064279; E-R9501; SWOG-9515
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation therapy (Active Comparator): Radiation therapy - 60 Gy in 6 weeks (2 Gy once a day, 5 x a week)
  Interventions: Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy
- Radiation therapy plus cisplatin (Experimental): Radiation therapy - 60 Gy in 6 weeks (2 Gy once a day, 5 x a week) plus Cisplatin-100 mg/m2 i.v. on days 1,22 and 43 with radiation therapy.
  Interventions: Drug: chemotherapy; Drug: cisplatin; Radiation: low-LET cobalt-60 gamma ray therapy; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Drug: chemotherapy
  Arms: Radiation therapy plus cisplatin
Drug: cisplatin
  Arms: Radiation therapy plus cisplatin
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether radiation therapy plus cisplatin is more effective than radiation therapy alone in treating patients with head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy plus cisplatin with radiation therapy alone in treating patients with head and neck cancer that has been removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate locoregional control rates, patterns of first failure, and overall and disease-free survival in patients with advanced squamous cell carcinoma of the head and neck at high risk of locoregional recurrence who are treated postoperatively with concurrent cisplatin and radiotherapy. II. Compare the toxicity of concurrent chemoradiotherapy vs. radiotherapy alone in the postoperative setting.

OUTLINE: Randomized study. Arm I: Radiotherapy. Involved-field irradiation using Co60, 1-6 MV photons, or electrons. Arm II: Radiotherapy plus Single-Agent Chemotherapy. Irradiation as in Arm I; plus Cisplatin, CDDP, NSC-119875.

PROJECTED ACCRUAL: 438 patients will be entered over approximately 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven squamous cell carcinoma of one of the following sites: Hypopharynx Larynx Oral cavity Oropharynx At least 1 of the following high-risk factors required: Histologic extracapsular nodal extension Histologic involvement of 2 or more regional lymph nodes Microscopically positive mucosal margins Complete resection of all visible and palpable disease Therapy must begin within 8 weeks of tumor-related surgery Bilateral resections may or may not be performed simultaneously Eligibility window begins with first definitive surgery Neck dissection not required for T4 N0, truly midline supraglottic tumors No tumors of the lip, nasopharynx, or sinuses No synchronous or concurrent head and neck tumors No evidence of distant metastasis Concurrent registration on Fixed Tumor Repository Study allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60%-100% Hematopoietic: WBC at least 3,500 Platelets at least 100,000 Hepatic: Not specified Renal: Creatinine clearance greater than 50 mL/min Other: No medical contraindication to protocol therapy No second malignancy within 5 years No pregnant or nursing women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to head and neck region Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 1995-09; Primary Completion 2002-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay S. Cooper, MD, FACR, FACRO, Study Chair — NYU Langone Health; James N. Endicott, MD, PA, Study Chair — H. Lee Moffitt Cancer Center and Research Institute; Julie A. Kish, MD, FACP, Study Chair — Josephine Ford Cancer Center
Locations (23):
- United States (22):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Background] Schumaker L, Nikitakis N, Goloubeva O, Tan M, Taylor R, Cullen KJ. Elevated expression of glutathione S-transferase pi and p53 confers poor prognosis in head and neck cancer patients treated with chemoradiotherapy but not radiotherapy alone. Clin Cancer Res. 2008 Sep 15;14(18):5877-83. doi: 10.1158/1078-0432.CCR-08-0998. PMID 18794100
- [Background] Bernier J, Cooper JS, Pajak TF, van Glabbeke M, Bourhis J, Forastiere A, Ozsahin EM, Jacobs JR, Jassem J, Ang KK, Lefebvre JL. Defining risk levels in locally advanced head and neck cancers: a comparative analysis of concurrent postoperative radiation plus chemotherapy trials of the EORTC (#22931) and RTOG (# 9501). Head Neck. 2005 Oct;27(10):843-50. doi: 10.1002/hed.20279. PMID 16161069
- [Result] Cooper JS, Zhang Q, Pajak TF, Forastiere AA, Jacobs J, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Lustig R, Ensley JF, Thorstad W, Schultz CJ, Yom SS, Ang KK. Long-term follow-up of the RTOG 9501/intergroup phase III trial: postoperative concurrent radiation therapy and chemotherapy in high-risk squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):1198-205. doi: 10.1016/j.ijrobp.2012.05.008. Epub 2012 Jun 30. PMID 22749632
- [Result] Cooper JS, Pajak TF, Forastiere AA, et al.: Long-term survival results of a phase III intergroup trial (RTOG 95-01) of surgery followed by radiotherapy vs. radiochemotherapy for resectable high risk squamous cell carcinoma of the head and neck. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-25, S14-5, 2006.
- [Result] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Result] Cooper JS, Pajak TF, Forastiere AA, et al.: Postoperative concurrent radiochemotherapy in high-risk SCCA of the head and neck: initial report of RTOG 9501/intergroup phase III trial. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-903, 2002.
- [Result] Cooper JS, Pajak TF, Forastiere AA, et al.: Patterns of failure for resected advanced head & neck cancer treated by concurrent chemotherapy and radiation therapy: an analysis of RTOG 9501/intergroup phase III trial. [Abstract] Int J Radiat Oncol Biol Phys 54(2 suppl 1): 2, 2002.